CLINICAL TRIAL: NCT01955577
Title: Vitamin D Supplement for Patients With Tibial Fracture Treated With an External Ring Fixator. A Prospective Randomized Double-blind Study.
Brief Title: Vitamin D Supplement for Patients With Tibial Fracture
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20130033
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Tibial Fracture
Keywords: Vitamin D deficiency; Ring fixator; Tibial fracture
MeSH Terms: conditions — Tibial Fractures; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 cholecalciferol (Experimental): 1000IU x3 daily in a period of 14 days. After 14 days 1000IU x 1 daily.
  Interventions: Drug: Vitamin D3 cholecalciferol
- Placebo orally everyday (Placebo Comparator): One placebo pill x3 daily in a period of 14 days. After 14 days x1 placebo pill daily.
  Interventions: Drug: Placebo orally everyday

INTERVENTIONS:
Drug: Placebo orally everyday
  Arms: Placebo orally everyday
Drug: Vitamin D3 cholecalciferol
  Arms: Vitamin D3 cholecalciferol

SUMMARY:
The purpose is to study:

1. the frequency of vitamin D deficiency at patients with tibial fracture treated with an external ring fixator
2. if vitamin D supplement facilitates fracture healing
3. a possible relation between vitamin D deficiency and the risk of complications and the time of fracture healing

DETAILED DESCRIPTION:
External ring fixator is a widespread and well-known method to treate complex tibial fractures. The effect of treating proximal and distal intra-articulatio tibial fractures has been positive until now.

Complications such as malunions, nonunions, re-fractures and extended time of ring fixation will occur in 5-10% of all tibial fractures in patients treated with ring fixator. Factors like trauma of soft tissue, smoking and compromised afflux of blood are associated with a higher frequency of nonunion.

It has been documented that elderly people with hypovitaminosis D have a higher risk of being affected by osteoporosis and fractures. Furthermore, there is a possible association between the severity of fracture and hypovitaminosis. The time of fracture healing is also extended compared to fractures in patients who are not affected by osteoporosis.

Until now research has not shown whether the fracture healing process is influenzed by vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tibial fracture
* A written signed statement of consent
* All potential patients primary with osteosynthesis Iliazov

Exclusion Criteria:

* Tumours in bone
* Metastases to bone marrow
* Chronic renal disease
* Drug abuse
* Abuse of alcohol (>21 drinks a week for men and > 14 drinks a week for women)
* Morbus Cushing disease
* Glandulae thyroid disease
* Pregnancy
* Chronic steroid therapy
* Hepatic insufficiency
* Sarcoidosis, tuberculosis or silocosis
* Patients under 18 years
* Inability to take medicine
* Adverse effects of vitamin D or allergic to vitamin D

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time of fracture healing | 20 weeks
  Time of fracture healing, i.e. time from osteosynthesis until fracture healing is clinically and radiologically registered.

SECONDARY OUTCOMES:
Vitamin D receptor DNA | 20 weeks
  A DNA blood sample will be taken in order to analyse how the skeleton reacts on vitamin D supplement.
Complications | 20 weeks
  Registration of possible complications, i.e. nonunion, malunion, number of check-ups, infections, re-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tine L. Bennedsen, M.D., Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Region Northern Jutland, Denmark